CLINICAL TRIAL: NCT00638482
Title: Pharmacodynamic Evaluation of the ANTICALCIURIC Effect of Hydrochlorothiazide in Dent's Disease
Brief Title: Dose-Dependent Effect of Thiazide in Dent's Disease Hypercalciuria
Acronym: DESY
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: terminated
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Saliha.DJANE, Department Clinical Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P011114; AOM 1093
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2008-03-19 (Estimated); Status verified 2003-07

CONDITIONS: Dent's Disease; Nephrolithiasis
Keywords: Dent's disease; Nephrolithiasis; clinical trial; thiazides
MeSH Terms: conditions — Dent Disease; Nephrolithiasis | interventions — Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Hydrochlorothiazide
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Hydrochlorothiazide — Hydrochlorothiazide

SUMMARY:
Intrarenal calcifications (nephrocalcinosis) is present in Dent's disease and likely contribute to progression toward renal failure. In order to prevent this complication it is usually proposed to treat affected patients during childhood with high doses of thiazides.

DETAILED DESCRIPTION:
Intrarenal calcifications (nephrocalcinosis) is present in Dent's disease and likely contribute to progression toward renal failure. In order to prevent this complication it is usually proposed to treat affected patients during childhood with high doses of thiazides. Indeed, this class of diuretics is used for years to treat hypertension, can lower urinary calcium excretion. However the doses usually used are high, are known to be associated with adverse events such as severe potassium depletion, decrease in blood pressure and dehydration. The purpose of the study was to test whether lower dose of thiazides would be better tolerated, with similar efficacy to lower urinary calcium excretion, as previously demonstrated in other indication such as treatment of hypertension.

Patient recruitment and clinical evaluation Eight subjects with genetically proven Dent's disease were recruited through a French nationwide network for tubulopathies and were enrolled between July 2003 and December 2005.

All patients met at least three standard criteria for the disease including hypercalciuria, low molecular weight proteinuria and one of the following disorders: nephrocalcinosis, nephrolithiasis, renal failure, aminoaciduria, glucosuria, renal phosphate wasting, or familial history of Dent's disease. The disease was confirmed in all patients by direct sequencing of the CLCN5 gene according to Lloyd et al. (25) Patients presenting hyponatremia (< 135 mM), hypokalaemia (< 3.3 mM), severe fanconi syndrome, or chronic renal failure (GFR estimated with the Schwartz formula < 30 mL.min-1.1.73m-2) were excluded from the study.

The protocol was approved by the "comité de protection des personnes" (Paris, Hôtel Dieu) and all subjects and/or their parents gave written informed consent for the participation in the study.

Sodium restriction test Because a renal loss of sodium was reported in the disease, the pharmacological study was preceded by a sodium restriction test involving NaCl intake equivalent to 0.3 mmol/kg BW) and an age-adjusted calcium intake of 1200-1500 mg/day, to assess the tolerance to sodium depletion and its effect on calcium excretion. Sodium restriction was stopped after 5 days or when 24h urinary sodium excretion matched theoretical salt intake. Blood and urine samples were taken in the morning, two hours after a light calcium-free breakfast and after a 30 minute rest in the supine position on the first and last days of the low sodium diet determining electrolytes, plasma proteins, hematocrit, and plasma renin and aldosterone concentrations.

PHARMACOLOGICAL STUDY After completion of the sodium restriction test, the seven remaining patients entered a three-period, forced titration sequential open-label trial. They were instructed to follow normal sodium, isocaloric diet, with an age-adjusted calcium intake of 1200 to 1500 mg/d. One patient had a tendency to hypokalaemia (3.3 mM), requiring potassium chloride salt supplementation before entering the trial.

After a one month run-in phase, the patients received sequentially a low dose (6.25 mg/day), an intermediate dose (12.5 mg/day), and a high dose (25 mg/day) of hydrochlorothiazide (HCTZ), each dose being administered for a period of two months. Amiloride (5 mg/day) was started at the beginning of the study, and continued throughout the sequential trial to reduce the risk of HCTZ-induced hypokalaemia. For safety reasons, two patients did not receive the last 25 mg dose of HCTZ because of a body weight (BW) < 25 kg. The last HCTZ dose was followed by a one month withdrawal period (phase E).

Clinical (blood pressure and BW), biological and hormonal evaluations were conducted at baseline and at the end of each treatment period, between 9:00 and 10:00 hours, two hours after a light calcium-free breakfast and a one hour-rest in a reclined position. At the end of the baseline and washout periods and each treatment period, two successive 24-h urine collections were obtained, and a morning spot urine sample was collected on the day of investigation for measurements of urine electrolytes (Na, K, calcium) and creatinine. Hematocrit, and electrolyte, creatinine, proteins, renin and aldosterone concentrations were measured in blood samples. Additionally, Blood Pressure, Body Weight and biological tolerance was assessed 15 days after each increase in the HCTZ dose.

Analytical methods Methods for the determination of plasma sodium, potassium, creatinine, magnesium, PTH, 25-OH vitamin D, renin, aldosterone and calcitriol levels have been described elsewhere.

Statistical Methods The effects of sodium restriction and HCTZ on clinical and biological markers were first evaluated by Friedman's tests. If a global time-effect was significant, the change between baseline and the last measurement of the treatment period was tested by a Wilcoxon's paired test. All data are expressed as median range [minimum; maximum], except otherwise specified. Values of 24h-urine collection of each period used for analyses were mean of the measurements made on the two consecutive daily collections. Values for a given 24-h collection were excluded from analysis if the creatinine excretion on that collection varied by more than 15% or the sodium excretion varied by more than 25% from the mean of values for other collections by that patient.

All analyses were carried out using SAS Statistical Software (Version 8.2, Cary, NC, USA) and STATVIEW(SAS Institute Inc., Cary NC) and a p value of less than 0.05 was considered to be significant.

ELIGIBILITY:
Inclusion Criteria:

* Children > 3 yrs old who met at least three standard criteria for Dent's disease including hypercalciuria, low molecular weight proteinuria and one of the following disorders: nephrocalcinosis, nephrolithiasis, renal failure, aminoaciduria, glucosuria, renal phosphate wasting, or familial history of Dent's disease.
* Dent's Disease confirmed by direct sequencing of the CLCN5 gene according to Lloyd et al.

Exclusion Criteria:

* Patients presenting hyponatremia (< 135 mM), hypokalaemia (< 3.3 mM), severe fanconi syndrome, or chronic renal failure (GFR estimated with the Schwartz formula < 30 mL.min-1.1.73m-2) were excluded from the study.
* Overt renal loss of sodium
* Inability to adapt to severe sodium restriction

Ages: 3 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2003-07; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
to investigate the dose-dependent benefit/risk ratio of low (6.25 mg/day), intermediate (12.5 mg/day) and high (25 mg/day) doses of hydrochlorothiazide | at the end of the baseline initial and final washout periods (one month each) and at the end of each two-months duration treatment period,

SECONDARY OUTCOMES:
clinical events (cramps, symptomatic dehydration, acute weight loss) | at least two times overall the study, at J15 and at the end of each period.
Biological : acute renal failure (estimated GFR), hypokalemia, hyperkalemia, hyponatremia, biological signs of extra cellular dehydration (protides, hematocrit, plasma active renin, plasma aldosterone) | at least two times overall the study, at J15 and at the end of each period.

CONTACTS AND LOCATIONS:
Overall Officials: Anne BLANCHARD, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Centre d'investigation clinique HOPITAL GEORGE POMPIDOU, Paris, France

REFERENCES:
- [Derived] Blanchard A, Vargas-Poussou R, Peyrard S, Mogenet A, Baudouin V, Boudailliez B, Charbit M, Deschesnes G, Ezzhair N, Loirat C, Macher MA, Niaudet P, Azizi M. Effect of hydrochlorothiazide on urinary calcium excretion in dent disease: an uncontrolled trial. Am J Kidney Dis. 2008 Dec;52(6):1084-95. doi: 10.1053/j.ajkd.2008.08.021. Epub 2008 Oct 30. PMID 18976849